CLINICAL TRIAL: NCT05651529
Title: Does Oral Intake of Beta-hydroxybutyrate Decrease Left Ventricular End-systolic Volume at Cardiac Magnetic Resonance in Patients With Heart Failure Compared to Carbohydrate Placebo?
Brief Title: Acute Oral Ketones or Carbohydrate Supplement Modify Heart Function in Heart Failure?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Nestlé Health Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2023-4720
Record Dates: First submitted 2022-11-29; First posted 2022-12-15 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure
Keywords: Ketones; Heart
MeSH Terms: conditions — Heart Failure; Ketosis | interventions — Postprandial Period

STUDY DESIGN:
Intervention Model Description: Crossover Assignment, Each participant will have to do the 2 Acute supplementation interventions
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple (Participant, Investigator, Outcomes Assessor) Investigators, participants and outcome assessors will be fully blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketone (Active Comparator)
  Interventions: Dietary Supplement: exogenous ketone salt supplement
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: exogenous carbohydrate supplement

INTERVENTIONS:
Dietary Supplement: exogenous ketone salt supplement — Dietary Supplement: Fasting water and with exogenous ketone salt supplement. Participants will have to take 1 doses of supplement 30 minutes before the scan.
  Other Names: Post-Prandial with exogenous ketone salt supplement
  Arms: Ketone
Dietary Supplement: exogenous carbohydrate supplement — Dietary Supplement: Fasting water and with exogenous carbohydrate supplement. Participants will have to take 1 doses of supplement 30 minutes before the scan.
  Other Names: Post-Prandial with exogenous carbohydrate supplement
  Arms: Placebo

SUMMARY:
Does oral intake of exogenous ketone salt improve heart function measured by cardiac MRI in heart failure compared to oral intake of a carbohydrate placebo?

DETAILED DESCRIPTION:
This study will help to quantify heart and kidney ketone uptake with or without an exogenous ketone salt in heart failure condition.

Participants will have 2 different cardiac MRI to perform:

1. Fasting with exogenous ketone salt supplement
2. Fasting with exogenous carbohydrate supplement

ELIGIBILITY:
Inclusion Criteria:

* Patients with heart failure with left ventricle ejection fraction of 40%
* Heart failure of ischemic or dilated etiology
* Ambulatory patient with a NYHA functional class of II-III;
* Stable symptoms and no change in medical therapy in the last month.

Exclusion Criteria:

* Diabetes
* Patients treated with any SGLT2i;
* Chronic kidney disease
* Acute coronary syndrome in the last 3 months;
* Use of parenteral inotropic agents;
* Persistent or permanent atrial fibrillation or atrial flutter;
* Presence of pacemaker or defibrillator;
* Medical condition that causes malabsorption of the test material;
* Under ketogenic diet, or using exogenous ketone supplements
* Use of nicotinamide adenine dinucleotide (NAD) precursor supplements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-12-16 (Actual); Primary Completion 2025-12-16 (Actual); Study Completion 2025-12-16 (Actual)

PRIMARY OUTCOMES:
Left ventricle ejection fraction by cardiac MRI under acute intake of exogenous ketone salt compared with exogenous carbohydrate placebo in heart failure patients. | 15 minutes
  Measure by Cardiac MR in pourcentage between diastolic and systolic volume in millimeter

SECONDARY OUTCOMES:
Right ventricle ejection fraction by cardiac MRI after intake supplement in heart failure patients. | 15 minutes
  Measure by Cardiac MR in pourcentage between diastolic and systolic volume in millimeter
Ventricle volume by cardiac MRI after intake supplement in heart failure patients. | 15 minutes
  Measure by Cardiac MR in millimeter
Cardiac output by cardiac MRI after intake supplement in heart failure patients. | 15 minutes
  Measure by Cardiac MR in liter per minute
Effects of supplement on serum biomarkers | 60 minutes
  Concentration of lactate (mmol/L)
Effects of supplement on serum biomarkers | 60 minutes
  Concentration sodium (mEq/L)
Effects of supplement on serum biomarkers | 60 minutes
  Concentration of N-terminal pro-B-type natriuretic peptide (NT-proBNP) (pg/ml)
Effects of supplement on serum biomarkers | 60 minutes
  Concentration of Beta-Hydroxybutyrate (mmol/L)
Effects of supplement on serum biomarkers | 60 minutes
  Concentration of glucose (mmol/L)
Effects of supplement on serum biomarkers | 60 minutes
  Concentration of insulin (IU)
Effects of supplement on the blood pressure of heart failure patients | 60 minutes
  Measure the blood pressure in systole and diastole in mm Hg
Effects of supplement on the heart rate of heart failure patients | 60 minutes
  Measure the heart rate in beat per minute

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Centre Hospitalier Universitaire de Sherbrooke, departement de cardiologie, Sherbrooke, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, departement de médecine, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Undecided